CLINICAL TRIAL: NCT02536976
Title: A Clinical Trial of Mirabegron for Overactive Bladder Symptoms in Patients With Parkinson Disease and Impaired Cognition
Brief Title: Mirabegron in Parkinson Disease and Impaired Cognition
Acronym: MICT-PD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 04412-15-A
Record Dates: First submitted 2015-08-28; First posted 2015-09-01 (Estimated); Results first posted 2019-05-08 (Actual); Last update posted 2019-05-08 (Actual); Status verified 2017-11

CONDITIONS: Parkinson Disease; Overactive Bladder; Impaired Cognition
Keywords: mirabegron
MeSH Terms: conditions — Parkinson Disease; Urinary Bladder, Overactive; Cognition Disorders | interventions — mirabegron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active treatment (Experimental): mirabegron
  Interventions: Drug: mirabegron
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: mirabegron
  Other Names: Myrbetriq
  Arms: Active treatment
Drug: Placebo
  Arms: Placebo

SUMMARY:
There is a high prevalence of OAB symptoms among patients with Parkinson's disease and a lack of pharmacotherapies with an acceptable side effect profile. Specifically, available anticholinergic medications have a high risk of cognitive side-effects, which preclude their use in PD patients with CI. PD can also cause a number of non-motor symptoms that are likely to be adversely affected by the currently available anticholinergic agents. Mirabegron is the first pharmacologic treatment which may not exacerbate CI, constipation, orthostatic hypotension (OH), somnolence, and dry mouth in PD.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Aged 25-80 at screening. Subjects older than 80 will be allowed at the discretion of the PI.
2. Ambulatory (defined as able to ambulate at least 10 meters, with or without assistance).
3. Clinical Diagnosis of PD based on the United Kingdom Brain Bank diagnostic criteria for PD.
4. At baseline visit (Visit 2) patients must have:

   * At least 8 micturitions per 24 hours and
   * At least 3 urgency episodes per 3-day diary.
5. A MoCA score between 19 and 28 (inclusive) at screening. For those on cognitive enhancers (donepezil, rivastigmine, memantine, galantamine) a MoCA score between 19 and 29 (inclusive) at screening.
6. Provide informed consent to participate in the study and understand that they may withdraw their consent at any time without prejudice to their future medical care.
7. Be cognitively capable, in the opinion of investigator, to understand and provide such informed consent.
8. Be cognitively capable to complete the required questionnaires and assessments, OR have a care partner who is willing and capable to assist them in the completion of these tasks.
9. Be on a stable regimen of antiparkinson's medications at least 30 days prior to screening, and be expected to remain on a stable dose for the duration of the study.
10. If taking cognitive enhancers (donepezil, rivastigmine, memantine, galantamine), must be on stable dose at least 30 days prior to screening, and be expected to remain on a stable dose for the duration of the study.

EXCLUSION CRITERIA:

1. Known or suspected alcohol or substance abuse in the preceding 12 months.
2. Women who are pregnant or breastfeeding.
3. Women of childbearing potential (WOCP) who are not using at least one method of contraception.
4. Patients with severe renal impairment (CLcr ≤ 29 mL/min, or eGFR ≤ 29 mL/min/1.73 m2), or moderate or severe hepatic impairment (Child-Pugh classes B or C).
5. Patients with bladder outlet obstruction (BOO) that, in the opinion of the study urologist, would expose them to risk of urinary retention during treatment with mirabegron.
6. Patients treated with drugs metabolized by the CYP2D6 pathway.
7. Patients with supine systolic blood pressure (SBP) ≥ 180 mm Hg, or diastolic blood pressure (DBP) ≥ 110 mm Hg.
8. Clinically significant, uncontrolled cardiac arrhythmia, unstable angina, congestive heart failure (NYHA Class 3 or 4), or history of myocardial infarction in the preceding 2 years.
9. History of cancer in the preceding 2 years other than successfully treated, non-metastatic, squamous cell or basal cell carcinoma, or cervical cancer in situ.
10. Any major urological procedure in the preceding 90 days.
11. Any major surgical procedure in the preceding 30 days.
12. Previously treated with mirabegron within 60 days prior to the baseline visit (Visit 2), or previously having failed treatment with mirabegron regardless of duration and timing of treatment.
13. Current or previous, within the 60 days preceding the baseline visit (Visit 2), treatment with antimuscarinic agents for OAB symptoms; and, willingness to not use antimuscarinic agents for the duration of the study.
14. Currently receiving any other investigational drug or having received an investigational drug within the 60 days preceding the baseline visit (Visit 2).
15. Any condition or laboratory test result, which, in the opinion of the Investigator or the Study Urologist, might result in an increased risk to the patient, or would affect their participation in the study.
16. Any patient who, in the opinion of the Investigator, is not a good candidate for the study or will not be able to follow study procedures.

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-12; Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sotirios A Parashos, MD, PhD, Principal Investigator — Struthers Parkinson's Center
Locations (1):
- Struthers Parkinson's Center, Golden Valley, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited in a single site from an ambulatory patient population of a dedicated Parkinson's Disease Center. First participant was screened in 12/2015 and the last participant completed the study in January 2018
Pre-assignment Details: 17 participants signed the ICF. There were 10 screen failures. 7 participants enrolled. 2 participants withdrew consent before starting study drug, and 1 was terminated during the placebo run-in phase due to unrelated failing health. 4 participants completed all study activities.
Groups:
- Active Treatment: Participants received 1 daily placebo tablet matching 25 mg tablets of mirabegron for 2 weeks , followed by 1 daily 25 mg tablet of mirabegron for 2 weeks, followed by 2 daily 25 mg tablets of mirabegron for 10 weeks.
- Placebo: Participants received 1 daily placebo tablet matching 25 mg tablets of mirabegron for 4 weeks , followed by 2 daily placebo tablets matching 25 mg tablets of mirabegron for 10 weeks.
Period: Overall Study
Arm/Group | Active Treatment | Placebo
Started | 3 (2 weeks single blind placebo run-in) | 2 (2 weeks single blind placebo run-in. 1 participant terminated due to unrelated failing health)
Randomization | 3 (2 weeks double blind mirabegron) | 1 (2 weeks double blind placebo matching mirabegron)
Dose Escalation and Maintenance | 3 (10 weeks double blind mirabegron) | 1 (10 weeks double blind placebo matching mirabegron)
Washout | 3 | 1
Completed | 3 | 1
Not Completed | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Active Treatment: 2 weeks single blind placebo followed by 2 weeks double blind 25 mg mirabegron, followed by 10 weeks double blind 50 mg mirabegron
- Placebo: 2 weeks single blind placebo followed by 2 weeks double blind placebo matching 25 mg mirabegron, followed by 10 weeks double blind 50 mg mirabegron
- Total: Total of all reporting groups
Arm/Group | Active Treatment | Placebo | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 0 | 2
  >=65 years | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 1 | 0 | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in Montreal Cognitive Assessment Total Score
Description: Change in Montreal Cognitive Assessment Total Score between week 2 and week 14. The Montreal Cognitive Assessment is a screening tool for global cognitive function with a total score ranging from 0 to 30 units on a scale, with higher score indicating better cognitive global function. Normal range is 26 thru 30.
Time Frame: From Week 2 to Week 14
Measure: Mean (Full Range); unit: units on a scale
Groups:
- Active Treatment: Due to sample size formal statistics were not performed. Observations tabulated below:
  Subject ID 8801 8814 8816 Change +2 +2 -1
- Placebo: Due to sample size formal statistics were not performed. Observations tabulated below:
  Subject ID 8805 Change +2
Arm/Group | Active Treatment | Placebo
Number analyzed (Participants) | 3 | 1
units on a scale | 1.5 [-1 to 2] | 2 [2 to 2]

2. Secondary Outcome: Change in Overactive Bladder Questionnaire Subscale Scores
Description: The Overactive Bladder Questionnaire (OABQ) is a 33-item, self-administered instrument that contains a symptom bother scale (8 items) and a health-related quality of life (HRQL) scale (25 items), pertaining to OAB symptoms impact on HRQL. Symptom bother score ranges from 0-100 with higher scores indicating greater severity of symptoms. The HRQL score ranges from 0-100 with higher scores indicating better quality of life.
Time Frame: From Week 2 to Week 14
Measure: Mean (Full Range); unit: units on a scale
Groups:
- Active: Participants receiving active treatment
- Placebo: Participants receiving placebo treatment
Arm/Group | Active | Placebo
Number analyzed (Participants) | 3 | 1
units on a scale
  Symptom Severity | -13.3 [-25 to 5] | 12.5 [12.5 to 12.5]
  HRQL | 13.7 [0 to 25] | 5 [5 to 5]

3. Secondary Outcome: Change in Unified Parkinson's Disease Rating Scale
Description: The UPDRS assesses motor and functional abilities of the subjects as it pertains to Parkinson's disease. The total UPDRS score (range 0-199; defined for this study as the sum of Parts I, II, III, and IV (I-Mentation, behavior, and mood section (4 items; range 0-16); II-Activities of Daily Living (ADL; 13 items; range 0-52); III-motor section (27 items; range 0-108) and IV-complications section; 11 items; range 0-23) will be completed by history and examination. Higher scores indicate greater severity of Parkinson's disease symptoms.
Time Frame: From Week 2 to Week 14
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Active | Placebo
Number analyzed (Participants) | 3 | 1
units on a scale | -5.3 [-16 to 6] | -9 [-9 to -9]

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | Active Treatment | Placebo
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 0/3 | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Treatment (N=3) | Placebo (N=2)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
headache (Nervous system disorders) | 0 (0) | 1 (1)
upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
cognitive dysfunction (Nervous system disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Study closed before reaching target enrollment. Due to the small number of participants enrolled no statistical analysis was performed, therefore no conclusions can be obtained.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-29): https://cdn.clinicaltrials.gov/large-docs/76/NCT02536976/Prot_SAP_000.pdf